CLINICAL TRIAL: NCT00378755
Title: Sequential VAD (Vincristine, Adriamycin, Dexamethasone) and VTD (Velcade, Thalidomide, Dexamethasone) Induction Followed by HDT With ASCT and Maintenance Treatment With Velcade for Newly Diagnosed MM
Brief Title: Sequential VAD and VTD Followed by HDT With ASCT and Velcade Maintenance for NDMM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean Multiple Myeloma Working Party (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMM51; 26866138MMY2028
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2006-09-22 (Estimated); Status verified 2006-09

CONDITIONS: Multiple Myeloma
Keywords: velcade; myeloma; VAD regimen; Transplantation, Autologous
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib

INTERVENTIONS:
Drug: velcade

SUMMARY:
1. Primary Objective To assess the response rate of sequential VAD (Vincristine, Adriamycin, Dexamethasone) and VTD (Velcade, Thalidomide, Dexamethasone) induction therapy as a first line treatment for the patients with multiple myeloma
2. Secondary Objectives

   1. To assess the progression free survival, duration of response, and overall survival of patients given sequential VAD and VTD induction followed by high dose therapy with autologous stem cell transplantation and maintenance treatment with Velcade
   2. To assess the toxicities of sequential VAD and VTD induction chemotherapy, high dose therapy with autologous stem cell transplantation, and of maintenance treatment with Velcade.

DETAILED DESCRIPTION:
1. Overview of study design

   This study aims to assess the efficacy and toxicities of sequential VAD and VTD induction followed by high dose therapy with autologous stem cell transplantation and maintenance treatment with velcade as a first line treatment for the patients with multiple myeloma. This study will be conducted as an open, multi-center, single arm, prospective phase 2 study.
2. Sample size determination

   The expected response rate of sequential VAD and VTD induction chemotherapy as a first line treatment for the patients with multiple myeloma is 80%. By using Flemming's single stage design ( error: 0.05,  error : 0.2), 55 evaluable patients are needed to prove this hypothesis. If withdrawal rate is 10%, enrollment of total 62 patients will be needed.
3. Duration of the Study

One year of enrollment will be needed (2006.03.1-2007.02.28). At least 24 months of follow-up for the patients who are to be enrolled last time is needed.

ELIGIBILITY:
Inclusion Criteria:

* 1.Previously untreated newly diagnosed patients with MM (stage II-III) 2.Age < 65 3.Eastern Cooperative Oncology Group Performance Status 0-1 4.EF > 50%, FVC and FEV > 50%, DLCO >50% 5.Platelet count ≥ 100 x 109/L (pretreatment platelet transfusion is not allowed, while transfusion during the treatment is permitted), hemoglobin ≥ 8 g/dL (≥ 4.96 mol/L), Prior RBC transfusion or recombinant human erythropoietin use is allowed), absolute neutrophil count (ANC) ≥ 1.0 x 109/L 6.Adequate liver function (bilirubin < UNL(Upper Normal Limit) x 2 and ALT/AST < UNL x 3) 7.Adequate renal function (serum creatinine < UNL x 1.5 or creatine clearance > 60 ml/min) 8.Signed the informed consent, have the will and ability to follow the protocol

Exclusion Criteria:

* 1. History of allergic reaction attributable to compounds containing boron or mannitol 2. Known hypersensitivity to thalidomide or dexamethasone 3. Peripheral neuropathy or neuropathic pain Grade 2 or higher as defined by NCI CTCAE version 3 4. Uncontrolled or severe cardiovascular disease, including MI within 6 months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis 5. Acute severe infection requiring antibiotic therapy 6. Previous cancer history (except in situ carcinoma of cervix or basal cell cancer of skin) 7. Pregnancy or breastfeeding 8. Active ulcer detected by gastroscopy (gastroscopy is not routine in all patients, only to patients with symptoms of ulcer disease and/or history of previous ulcer therapy and/or physician's discretion) 9. Previous renal transplantation 10. Recurrent deep vein thrombosis or pulmonary embolism 11. Uncontrolled diabetes mellitus 12. Receipt of extensive radiation therapy within 4 weeks ((Extensive means RT to more than 2 anatomic sites).

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62
Dates: Start 2006-03; Study Completion 2008-07

PRIMARY OUTCOMES:
response rate of sequential VAD (Vincristine, Adriamycin, Dexamethasone) and VTD (Velcade, Thalidomide, Dexamethasone) induction therapy as a first line treatment for the patients with multiple myeloma

SECONDARY OUTCOMES:
the progression free survival
duration of response
overall survival
toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Soo Yoon, MD PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea